CLINICAL TRIAL: NCT05223569
Title: Home Monitoring of Diabetic Macular Edema
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021KYPJ099
Record Dates: First submitted 2022-01-22; First posted 2022-02-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-02

CONDITIONS: Macular Edema Due to Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home OCT monitoring model (Experimental): Participants will receive a home monitoring set, which includes a self-administrated OCT, and a self-administrated smartphone-based visual acuity tester. For each home service, participants will undergo the following:
  1. Smartphone-assisted online instruction provided by a virtual specialist
  2. Visual acuity self test using a smartphone
  3. Self-testing OCT imaging
  Interventions: Device: Home OCT monitoring model
- Hospital-based monitoring with a staff-administrated OCT (Active Comparator): Participants will be instructed to come back to the clinic to receive traditional OCT and VA examinations operated by the study coordinators every month.
  Interventions: Device: Hospital-based monitoring with a staff-administrated OCT

INTERVENTIONS:
Device: Home OCT monitoring model — A home monitoring set, which includes a self-administrated OCT, and a self-administrated smartphone-based visual acuity tester
  Arms: Home OCT monitoring model
Device: Hospital-based monitoring with a staff-administrated OCT — Participants come back to the clinic to receive traditional OCT and VA examinations operated by the study coordinators
  Arms: Hospital-based monitoring with a staff-administrated OCT

SUMMARY:
Diabetic macular edema (DME) is part of diabetic retinopathy (DR) and a leading cause of central visual loss in people with diabetes . Most patients require pharmacological inhibition using anti-vascular endothelial growth factor (VEGF) agents with multiple monitoring visits that include optical coherence tomography (OCT), visual acuity test, and multiple injections.The substantial visit frequency puts pressure on ophthalmic clinics, and can impose a tremendous burden on both patients and their caregivers. Therefore, self-service examination instruments that can be portable and fast-moving become the key for realizing tele-medicine. Recently, the investigators have developed a portable, self-administrated home OCT machine, which is designed for home-based OCT scanning and monitoring for patients with retinal diseases including DME, age related macular degeneration (AMD) and choroidal neovascularization (CNV) that require multiple anti-VEGF injections. The investigators have confirmed its image quality and validated the retinal thickness measurements obtained from this device by comparing with hospital OCT (staff-administrated and clinic-based).In this study, the investigators will conduct a randomized clinical trial (RCT) to compare the efficacy and cost-effectiveness of a home OCT monitoring model versus standard hospital care model for patients with diabetic macular edema who need anti-VEGF injections.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. Diagnosis of diabetic macular edema:

   * Type 1 or type 2 diabetes mellitus;
   * Center-involved macular edema;
3. Willing to receive anti-VEGF treatment;
4. Media clarity, pupillary dilation, and individual cooperation sufficient for adequate OCT examination;
5. Able to operate self-administratedhome OCT by themselves or with the help of family;
6. Travel time from home to hospital: within 2 hours driving.
7. Able and willing to provide informed consent.

Exclusion Criteria:

1. History of systemic anti-VEGF or pro-VEGF treatment within 4 months prior to randomization. (These drugs should not be used during the study);
2. History of corticosteroid treatment (intravitreal or peribulbar) at any time in the past 4 months;
3. History of macular laser photocoagulation in the past 4 months;
4. Macular edema due to reasons other than diabetes;
5. Coexisting ocular diseases that might alter visual acuity during the course of the study, such as retinal vein or artery occlusion, uveitis or other ocular inflammatory disease, neovascular glaucoma, etc.);
6. Hypertension (systolic blood pressure (BP) above 180 or diastolic BP above 110);
7. History of myocardial infarction, other acute cardiac event requiring hospitalization, stroke, transient ischemic attack, or treatment for acute congestive heart failure within 4 months prior to randomization;
8. Pregnant or lactating;
9. Currently participating in other clinical trials;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-03-03 (Actual); Primary Completion 2023-12-12 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Changes in visual acuity | 12 weeks
  Changes in visual acuity from baseline to 12 weeks adjusted for baseline visual acuity

SECONDARY OUTCOMES:
The costs of treatment | 12 weeks
  The Cost-effectiveness between the two monitoring models
Number of intravitreal injections | 12 weeks
  The number of intravitreal injections given per group
Gains or losses in visual acuity | 12 weeks
  The proportion of eyes with two- and three-line gains or losses in visual acuity
Central subfield thickness change as measured by optical coherence tomography | 12 weeks
  central subfield thickness and retinal volume as measured by OCT after 12 weeks
Number of visits | 12 weeks
  The number of visits during the study
Changes in visual acuity after 24 weeks | 24 weeks
  Changes in visual acuity from baseline to 24 weeks adjusted for baseline visual acuity
Changes in visual acuity after 48 weeks | 48 weeks
  Changes in visual acuity from baseline to 48 weeks adjusted for baseline visual acuity

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Han X, Scheetz J, Keel S, Liao C, Liu C, Jiang Y, Muller A, Meng W, He M. Development and Validation of a Smartphone-Based Visual Acuity Test (Vision at Home). Transl Vis Sci Technol. 2019 Aug 19;8(4):27. doi: 10.1167/tvst.8.4.27. eCollection 2019 Jul. PMID 31440424
- [Background] Maloca P, Hasler PW, Barthelmes D, Arnold P, Matthias M, Scholl HPN, Gerding H, Garweg J, Heeren T, Balaskas K, de Carvalho JER, Egan C, Tufail A, Zweifel SA. Safety and Feasibility of a Novel Sparse Optical Coherence Tomography Device for Patient-Delivered Retina Home Monitoring. Transl Vis Sci Technol. 2018 Jul 24;7(4):8. doi: 10.1167/tvst.7.4.8. eCollection 2018 Jul. PMID 30050725
- [Background] Weiss M, Sim DA, Herold T, Schumann RG, Liegl R, Kern C, Kreutzer T, Schiefelbein J, Rottmann M, Priglinger S, KortUEm KU. COMPLIANCE AND ADHERENCE OF PATIENTS WITH DIABETIC MACULAR EDEMA TO INTRAVITREAL ANTI-VASCULAR ENDOTHELIAL GROWTH FACTOR THERAPY IN DAILY PRACTICE. Retina. 2018 Dec;38(12):2293-2300. doi: 10.1097/IAE.0000000000001892. PMID 29068914
- [Background] Jusufbegovic D, Mugavin MO, Schaal S. EVOLUTION OF CONTROLLING DIABETIC RETINOPATHY: Changing Trends in the Management of Diabetic Macular Edema at a Single Institution Over the Past Decade. Retina. 2015 May;35(5):929-34. doi: 10.1097/IAE.0000000000000438. PMID 25590856